CLINICAL TRIAL: NCT06827639
Title: In-depth Characterization of Circulating and Infiltrating Immune Subsets and Tumor Cells in Cancer Patients.
Acronym: FUTURE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23-0388; 2023-A02198-37 (Registry Identifier: ID RCB)
Record Dates: First submitted 2024-08-28; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer; Urologic Cancer; Lung Cancer; Breast Cancer; Liver Cancer
Keywords: Tumor microenvironment; Immuno-phenotyping; Immunohistochemistry; Ex-vivo functional assays; circulating tumor DNA; Gene sinatures; Breast cancer; Head and neck cancer; Urologic cancer; Liver cancer; Colorectal and gastric cancer; Lung cancer; lymphoma; leukemia
MeSH Terms: conditions — Head and Neck Neoplasms; Urologic Neoplasms; Lung Neoplasms; Breast Neoplasms; Liver Neoplasms; Stomach Neoplasms; Lymphoma; Leukemia | interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples will be retained for phenotyping by flow cytometry, immune cells isolation for functional tests, nucleic acids extraction, cell freezing and storage, serum, plasma and PBMC preparation, freezing and storage
  * Fresh tissues from surgical resections will be obtained according to planned, standard medical practice. Remaining biological material only will be used and retained for tissue sample dissociation, ex vivo functional assays, tissue freezing or fixation and storage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1 - Patients with solid tumor undergoing surgery: Cohort 1 (patients with solid tumor undergoing surgery):
  * Head and neck cancer: up to 80 patients
  * Urologic cancer: up to 160 patients
  * Liver cancer: up to 80 patients
  * Colorectal and gastric cancer: up to 80 patients
  * Breast cancer: up to 80 patients
  A maximum of 3 visits are planned :
  * Screening visit for patient evaluation and inclusion/exclusion criteria review
  * Visit 1: For blood sampling specifically for the study
  * Visit 2: For tumor sampling and blood sampling if not done at Visit 1 Fresh solid tumor lesions and normal adjacent tissue will be macroscopically selected from the resected tumor material by a pathologist. Samples will be collected according to decision of May 3, 2017 establishing a list of researches as mentioned by article L1121-1, paragraph 2° of the French public Health code, and will therefore only concern blood samples, as well tissues collected during surgeries.
  The Screening visit and the Visit 1 can occur on the same day.
  Interventions: Procedure: blood collection; Procedure: tissue specimen collection
- Cohort 2 - Patients with solid tumor with anti-PD1/PD-L1 treatment and no surgery: * Lung cancer: up to 40 patients
  * Head and neck cancer: up to 40 patients a maximum of 3 visits are planned during this period:
  * A Screening visit for patient evaluation and inclusion/exclusion criteria review.
  * A Baseline visit (pre-treatment) visit for blood sampling specifically for the study
  * A post-treatment visit (after immunotherapy administration) for blood sampling specifically for the study The Screening and Baseline visits can occur on the same day.
  Interventions: Procedure: blood collection
- Cohort 3 - Patients with hematological malignancies: - Lymphoma and leukemia: up to 80 patients
  A maximum of 2 visits are planned during this period:
  * A Screening visit
  * Visit 1: for blood sampling specifically for the study The Screening visit and the Visit 1 could occur on the same day.
  Interventions: Procedure: blood collection

INTERVENTIONS:
Procedure: blood collection — Blood sampling is performed during Scrrening / visit 1 for patients enrolled in cohort 1, cohort 2 and cohort 3
Procedure: tissue specimen collection — In Cohort 1- patients with solid tumor undergoing surgery, fresh tissue specimen is collected during surgery
  Groups: Cohort 1 - Patients with solid tumor undergoing surgery

SUMMARY:
The aim of this study is to describe the tumor microenvironment of solid tumors and to understand the changes induced by anti-cancer treatments, particularly those developed by Innate Pharma. Innate Pharma is a biotechnology company which discovers and develops therapeutic antibodies that exploit the innate immune system to improve cancer treatment. Thanks to this study, it will be possible to correlate clinical and immunological characteristics with the patient's clinical features. The analyses generated will contribute to the design and improvement of innovative therapeutic antibodies acting on the immune system

DETAILED DESCRIPTION:
Rationale:

The purpose of this study is to characterize the tumor and immune contexture and its circulating counterpart in cancer patients and to understand changes induced by anti-cancer treatments. We will therefore be able to correlate clinical and immunological characteristics with patient clinical status. We expect that the data generated will be used as a decision-support tool for the design and evaluation of new or improved immunotherapy.

Study objectives:

* Primary objectives:
* Identification and functional characterization of circulating and infiltrating immune subsets and tumor cells in cancer patients.
* Discovery and preclinical evaluation of new therapeutic targets in oncology.

Secondary objectives:

* To evaluate and compare the frequency, phenotype and functionality of leukocytes subsets in the tumor microenvironment, tumor-adjacent tissue and in peripheral blood.
* To evaluate the expression of proteins targeted by therapeutic antibodies on circulating and tissue-resident cells in cancer patients.
* To assess the impact of anti-cancer treatments (including but not limited to therapeutic antibodies or chemotherapy) on the tumor and peripheral microenvironment (e.g. frequency and phenotype of leukocyte subsets; expression of targeted proteins or their ligands).
* To identify correlation between tumor biomarkers / blood biomarkers and biological or clinical characteristics of cancer patients as well as their clinical response to treatment.
* To characterize ex vivo the modes of action of several anti-cancer treatments.

Study Design:

During this study, patients will not receive any investigational product. Patients are included within their usual schedule of appointments with their surgeon or oncologist. Treatment strategy (surgery, chemotherapy, immunotherapy…) will vary from indication to indication and will not be impacted by participation to this study.

Screening and sampling Period

For patients with solid tumor undergoing surgery (cohort 1), a maximum of 3 visits are planned during this period:

* A Screening visit for patient evaluation and inclusion/exclusion criteria review
* Visit 1: For blood sampling specifically for the study;
* Visit 2: For tumor sampling and blood sampling if not done at Visit 1. Fresh solid tumor lesions and normal adjacent tissue will be macroscopically selected from the resected tumor material by a pathologist. Samples will be collected according to decision of May 3, 2017 establishing a list of researches as mentioned by article L1121-1, paragraph 2° of the French public Health code, and will therefore only concern blood samples, as well tissues collected during surgeries.

The Screening visit and the Visit 1 could occur on the same day.

For patients with solid tumor registered for anti-PD1/PD-L1-based treatment and not undergoing surgery (cohort 2), a maximum of 3 visits are planned during this period:

* A Screening visit for patient evaluation and inclusion/exclusion criteria review.
* A Baseline (pre-treatment) visit for blood sampling specifically for the study.
* A Post-treatment (after immunotherapy administration) for blood sampling specifically for the study.

The Screening and Baseline visits could occur on the same day.

For hematological malignancies (cohort 3), a maximum of 2 visits are planned during this period:

* A Screening visit;
* Visit 1: for blood sampling specifically for the study. The Screening visit and the Visit 1 could occur on the same day.

Target patient population:

Age ≥ 18 years with one of the following cancer indication:

* Lung cancer,
* Head and neck cancer,
* Urologic cancer,
* Liver cancer,
* Colorectal and gastric cancer,
* Breast cancer,
* Lymphoma and leukemia

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologic, cytologic or imaging confirmation of a malignancy in accordance with targeted indications
* Written informed consent signed from subject prior to performing any protocol-related procedures

Exclusion Criteria:

* Use of any investigational agent within 14 days prior first visit;
* Patient under guardianship/trusteeship or legally incapacitated person;
* Patient unable to understand read and/or sign an informed consent;
* Uncooperative or potentially non-compliant for the study or study procedures patient, or with foreseeable regular follow-up difficulties;
* Patient without Health insurance scheme or Universal Medical Coverage (CMU) or any equivalent scheme;
* Patients who are known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from hospitals in Assistance Public Hopitaux de Marseille : Nord, Conception and Timone
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of circulating and infiltrating tumor cells . | From screening to end of study at 8 weeks
  Caracterization of tumor cells immuno-phenotyping and gene signature.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic VELY, Dr, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hopital Timone enfants - plateforme d'Immunoprofiling, Marseille, France

IPD SHARING:
Plan to Share IPD: No